CLINICAL TRIAL: NCT01120197
Title: Study of Effect of Exercise on Health-related Quality of Life, Mobility and Balance in Osteoporotic Women With a History of Vertebral Fracture.
Brief Title: Study of Effect of Exercise With Osteoporosis and Vertebral Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 301.0
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: randomized controlled trial; osteoporosis; moderate-intensity circuit exercises; balance; health-related quality of life
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental): Exercise group with intervention
  Subjects in the intervention group must participate in a training course consisted of 24 sessions over 3 months. The exercises include aerobic, stretching, balance and functional training, i.e. circuit exercises focus been on: the prevention of falls and fractures, improving balance and coordination, improving posture, and informing subjects about risk factors for falls and for osteoporosis and fractures. A 3-hour session of information and supervision will be hold for the intervention group by the same physiotherapist who leads the training sessions. The focus is on body awareness and ergonomic advice in specific, daily-life situations (e.g. lifting/carrying, resting positions).
  Interventions: Other: Exercise group
- Control Group (Other): Control group with no intervention
  Subjects in the control group are asked to maintain their current lifestyle. No restrictions are placed on their exercise activities. The control group is followed for the same duration as the intervention group.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Exercise group — Weekly exercises
  Arms: Exercise group
Other: Control Group — No Intervention, control group only
  Arms: Control Group

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effectiveness for health-related quality of life (HRQOL) of a 3-month course of exercises for a group of postmenopausal women with osteoporosis who has at least one vertebral fracture versus a control group (undertaking their usual activities). The course of exercises is devised in accordance with methods recommended in "Rehabilitation treatment guidelines in postmenopausal and senile osteoporosis".

DETAILED DESCRIPTION:
Public health policies in most European countries are concerned with how to keep older people living independently with a qualitatively good life in the community as long as possible. Apart from its personal and human cost, osteoporosis is a major public health problem, which has an enormous social and economic impact. Osteoporosis(OP) is a common condition among older people,and a non-fatal condition that leads more to changes in the quality of life than to change in the length of life. Osteoporosis is a skeletal disorder characterized by decreased bone mass. The World Health Organization (WHO) Study Group on Osteoporosis has defined osteoporosis as "a hip BMD level of more than 2.5 SDs below the mean BMD for young, white, adult women". Using the WHO definition, approximately 30% of postmenopausal women have osteoporosis.

The most common consequences of osteoporosis are fractures. Furthermore the most common conditions associated with osteoporosis are back pain, limitations in physical functioning, and psychosocial impairment. Thus, the purpose of this study is to record the effect of the programme on mobility, balance, the disease-specific and generic health-related quality of life for women with osteoporosis and a history of vertebral fractures. The programme consist of a three-hour educational session and a three-month course of exercises in accordance with guidelines for women with an increased risk of falls and postmenopausal osteoporotic women with a history of fractures.

Our hypothesis that a three-month course of exercises and a three-hour lesson on how to cope with osteoporosis will have a significantly positive effect on the generic and disease-specific quality of life, as well as the balance and mobility, of elderly (≥60 years) women with postmenopausal osteoporosis and a history of vertebral fractures, both 3 months after the intervention and after one year.

The sample would be recruited from the Osteoporosis Outpatient clinic at the Ostfold Hospital, Norway and they their body mineral density (BMD) has been measured using Dual-Energy X-Ray Absorptiometry (DXA). The design of the study is a randomized controlled trial and the sample would be randomized to an intervention group or a control group.

Subjects in the control group are asked to maintain their current lifestyle. No restrictions are placed on their exercise activities. Subjects in the intervention group must participate in a training course consisted of 24 sessions over 3 months. The exercises include aerobic, stretching, balance and functional training, i.e. circuit exercises focus been on: the prevention of falls and fractures, improving balance and coordination, improving posture, and informing subjects about risk factors for falls and for osteoporosis and fractures.

A 3-hour session of information and supervision will be hold for the intervention group by the same physiotherapist who leads the training sessions. The focus is on body awareness and ergonomic advice in specific, daily-life situations (e.g. lifting/carrying, resting positions).

ELIGIBILITY:
Inclusion Criteria:

* women
* living at home
* ambulatory
* aged 60 or more
* clinical diagnosis of osteoporosis
* a history of vertebral fracture

Exclusion Criteria:

* recent vertebral fractures
* unable to complete the questionnaires
* major cognitive impairment (MMSE) ( MMS < 23 )

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-05; Primary Completion 2009-01 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, Professor, Study Director — Faculty of Health Science, University of Oslo, Norway
Locations (1):
- Ostfold Hospital Trust, Sarpsborg, Norway

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Group: Exercise Group: Subjects in the intervention group must participate in a training course consisted of 24 sessions over 3 months. The exercises include aerobic, stretching, balance and functional training, i.e. circuit exercises focus been on: the prevention of falls and fractures, improving balance and coordination, improving posture, and informing subjects about risk factors for falls and for osteoporosis and fractures. A 3-hour session of information and supervision will be hold for the intervention group by the same physiotherapist who leads the training sessions. The focus is on body awareness and ergonomic advice in specific, daily-life situations (e.g. lifting/carrying, resting positions).
  The intervention is in accordance with Rehabilitation treatment guidelines in postmenupausal and senile osteoporosis ( Bonaiuti et al. 2005).
- Control Group: Control group with no intervention
  Subjects in the control group are asked to maintain their current lifestyle. No restrictions are placed on their exercise activities
Period: Overall Study
Arm/Group | Exercise Group | Control Group
Started | 47 | 42
Completed | 38 | 32
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Exercise Group: : Subjects in the intervention group must participate in a training course consisted of 24 sessions over 3 months. The exercises include aerobic, stretching, balance and functional training, i.e. circuit exercises focus been on: the prevention of falls and fractures, improving balance and coordination, improving posture, and informing subjects about risk factors for falls and for osteoporosis and fractures. A 3-hour session of information and supervision will be hold for the intervention group by the same physiotherapist who leads the training sessions. The focus is on body awareness and ergonomic advice in specific, daily-life situations (e.g. lifting/carrying, resting positions).
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Control Group | Total
Number analyzed (Participants) | 47 | 42 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 47 | 42 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (5.9) | 72 (5.8) | 71.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 42 | 89
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Norway | 47 | 42 | 89

OUTCOME MEASURES:

1. Primary Outcome: Time Used to Walk 20 m at Maximal Speed.
Description: Times (measured in seconds) used walking at maximum speed for 20m indoors. No acceleration or deceleration phase used. The type of walking aids used during the test will be recorded. The participants walk as fast as possible wearing their ordinary shoes. The test perform once, the time measured with a stopwatch and the time used on 20 m will be recorded
Time Frame: At baseline, 3 and 12 months after the baseline
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Exercise Group: Subjects in the intervention group must participate in a training course consisted of 24 sessions over 3 months. The exercises include aerobic, stretching, balance and functional training, i.e. circuit exercises focus been on: the prevention of falls and fractures, improving balance and coordination, improving posture, and informing subjects about risk factors for falls and for osteoporosis and fractures. A 3-hour session of information and supervision will be hold for the intervention group by the same physiotherapist who leads the training sessions. The focus is on body awareness and ergonomic advice in specific, daily-life situations (e.g. lifting/carrying, resting positions).
- Control Group: Control group with no intervention
  Subjects in the control group are asked to maintain their current lifestyle. No restrictions are placed on their exercise activities. [We recommend specifying length of time they are followed]
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 47 | 42
Seconds
  Baseline | 14.9 (4.3) | 14.7 (3.5)
  3 months | 13.4 (4.1) | 15.2 (4.3)
  12 months | 13.8 (4.7) | 15.3 (4.7)

2. Secondary Outcome: Timed Up & Go Test (TUG)
Description: The subject will be instructed to rise from a chair with a seat height of 43 cm, walk 3 m, turn around, return and sit down again, wearing ordinary footwear and use customary walking aids if necessary.
Time Frame: At baseline, 3 and 12 months after the baseline.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 47 | 42
Seconds
  Baseline | 7.9 (2.6) | 8.3 (2.4)
  3 months | 7.5 (2.1) | 8.7 (2.8)
  12 months | 7.3 (2.1) | 8.5 (2.5)

3. Secondary Outcome: Functional Reach
Description: The maximum distance in centimetres that can be reached forward in a standing position while maintaining a fixed base of support. Subjects will be instructed to stand sideways against a wall in a natural position and stretch one arm forward level with the shoulder. The position of the third metacarpophalangeal (MCP) joint was taken as the zero point. With the body tilted forward as far as possible, the subjects continued to stretch the arm parallel to the ground.
  Amount of cm indicate better balance.
Time Frame: At baseline, 3 and 12 months after the baseline
Measure: Mean (Standard Deviation); unit: Centimetres
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 47 | 42
Centimetres
  Baseline | 26.1 (6.7) | 27.4 (6.3)
  3 months | 27.7 (6.5) | 25.2 (7.5)
  12 months | 27.1 (6.5) | 27.7 (5.4)

4. Secondary Outcome: QUALEFFO 41
Description: Quality of Life Questionnaire issued by the European Foundation for Osteoporosis (QUALEFFO-41), is a disease-specific questionnaire to be used by patients with vertebral fractures attributed to osteoporosis. QUALEFFO-41 is self-administered and contains questions in five domains: pain, ability to perform physical functions, social functioning, general health perception and mental performance. These five domains can be evaluated individually or be represented in a total score. All scores in all the domains are expressed in values ranging from 0-100, where 0 represents the best and 100 the worst. The total QALEFFO score is calculated as a sum of all answers to items and then linearly transformed on the scale 0-100.
  High scores indicate poor quality of life.
Time Frame: At baseline, 3 and 12 months after the baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 47 | 42
units on a scale
  Baseline | 31.8 (14.4) | 31.3 (13.3)
  3 months | 29.8 (14.3) | 31.5 (14.9)
  12 months | 28.7 (13.5) | 31.7 (14.8)

5. Secondary Outcome: General Health Questionnaire 20 (GHQ20).
Description: GHQ-20 is a generic instrument and registers distress and psychopathology. GHQ-20 is self-administered and the answers to each item may be treated as a "Likert Scale" and have weights assigned to each position (0-1-2-3) where 0 is no distress, and 3 is severe distress. This gives a possible range for the total GHQ-20 score of 0-60. Higher scores indicating poor qol.
Time Frame: At baseline, 3 and 12 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 47 | 42
units on a scale
  Baseline | 18.7 (8.8) | 20 (6.9)
  3 months | 15.1 (7) | 19.8 (7.4)
  12 months | 16.1 (7.1) | 19 (6.1)

6. Secondary Outcome: Falls-Efficacy Scale-International
Description: A 16- item self report or interview- based questionnaire assessing the fear of falling during basic and more demanding activities of daily living (Yardley et al. 2005). Each item is scored on a four point scale. Minimun score indicating low concern about falling is 16. The maximun score indication high concern about falling is 64.
Time Frame: Baseline, 3 months follow-up, 12 months follow up
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse events were systematically reported in the way that participants held log diaries after each exercise session (any adverse events: yes/no). Any adverse event would have been further investigated by the researchers.
Arm/Group | Exercise Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/42
Other Adverse Events (participants affected / at risk) | 0/47 | 0/42

LIMITATIONS AND CAVEATS:
The numbers in our study were relatively small, and some caution is required in interpretation. Additionally, it cannot be ruled out that participants have become aware of the treatment allocation, and this could potentially have biased the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No